CLINICAL TRIAL: NCT04661111
Title: Prospective, Monocentric, Study to Assess Efficacy and Safety of Hymovis® ONE (32 mg/4 ml) Intra-articular Injection in Active Patients Affected by Knee Overuse Syndrome
Brief Title: Efficacy and Safety of Hymovis ONE® (32mg/4ml) Intrarticular Injection in Active Patients With Knee Overuse Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQL2-15-01
Record Dates: First submitted 2020-03-02; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hymovis ONE Arm (Experimental): Hymovis® ONE (32 mg/4 ml) intra-articular mono injection. Patients will be followed during 12 months including 6 visits.
  Interventions: Device: Hymovis® ONE (32 mg/4 ml)

INTERVENTIONS:
Device: Hymovis® ONE (32 mg/4 ml) — Hymovis® ONE is a clear hydrogel. The conjugate compound is constituted by a partial hexadecylamide of hyaluronic acid, which is produced by a fermentation process. Hymovis® ONE is a CE-marked Class III Medical Device intended for intra-articular injection.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Hymovis® ONE (32 mg/4 ml) single intra-articular injection, in the management of pain caused by knee osteochondral lesions.

DETAILED DESCRIPTION:
There are no studies in literature up to now, that analyze the changes in knee pain and correlate this parameter with knee function and biomechanics, in regular casual sport player subject affected by knee overuse syndrome and underwent an intra-articular HA injection. The aim of this study is to evaluate efficacy and safety of Hymovis® ONE (32 mg/4 ml) single intra-articular injection, in the management of pain caused by knee osteochondral lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female higher than 18 and less or equal to 65 years of age
2. an active life-style, professional or regular casual sport player (people who plays sport or trains themselves at least 2-3 times per week).
3. diagnosis of knee osteoarthritis will be based upon a standing weight bearing knee X-ray at Screening or an X-ray performed within 6 months prior to screening. The radiograms must be classified as a Kellgren and Lawrence Grade I-III for osteoarthritis of the knee.
4. a knee VAS pain score, within 48 hours before the visit.
5. patients must have had all analgesic/anti-inflammatory drugs discontinued for 2 weeks prior to Baseline except for acetaminophen.

Exclusion Criteria:

1. Major injury to the contralateral knee or other weight-bearing joint if it would interfere with the study assessments.
2. Surgical procedure of the studied joint within the previous 12 months prior to Screening.
3. Ligament reconstruction in the target knee within 1 year
4. Inflammatory arthropathies such as rheumatoid arthritis, lupus, or psoriatic arthritis
5. Intra-articular or local peri-articular corticosteroid injections to the study joint/knee within the previous 3 months prior to screening or to any other joint (beside the study joint) or soft tissue area within the previous month prior to Screening.
6. Any corticosteroid within the previous month. Steroid inhalants are permitted if the patient has been on a stable regimen for the past month prior to Screening and remains on this regimen throughout the course of the trial.
7. Intra-articular hyaluronan in the studied joint within the previous 6 months prior to Screening.
8. History of allergic reaction to an intra-articular Hyaluronic acid injection
9. Use of glucosamine- or chondroitin sulfate-containing products unless the patient is on stable doses for at least 4 months prior to Screening and willing to remain on these stable doses throughout the course of the trial.
10. Patients with X-ray findings of acute fractures, severe loss of bone density, avascular necrosis and/or severe deformity.
11. Axial deviation of the lower limbs higher than 20 degrees in valgus or varus on standing X-ray.
12. Symptomatic osteoarthritis of either hip, contralateral knee or spine that may interfere with functional assessment of the signal knee.
13. Clinically significant medio-lateral and/or anterior-posterior instability.
14. Osteonecrosis of either knee.
15. If patients are receiving or performing physical therapy at Screening, this physical therapy regimen has not been stable during the one-month preceding Screening and the patient is not willing to maintain the same regimen throughout the course of the trial.
16. Patients with Kellgren-Lawrence Stage IV osteoarthritis of the knee (i.e.,in grade IV large osteophytes, marked narrowing, severe sclerosis, and definite deformity).
17. Hemiparesis of the lower limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
The efficacy of Hymovis® ONE (32 mg/4 ml) single intra-articular injection, in the management of pain caused by knee osteoarthritis due to overuse: KOOS questionnaire (Knee injury and Osteoarthritis Outcome Score) | Day 90 after baseline visit
  To demonstrate that a single intra-articular (i.a.) injection of Hymovis® ONE (32 mg/4 ml) decreases the difficulties in sport and recreational activity. The efficacy will be measured evaluating the improved knee function during sport and recreational activity through the fourth item (SP1-SP5) of the KOOS questionnaire, 90 days after injection. A five-point Likert scale(LK3 series) will be used to score each of the five KOOS questionnaire items (Symptoms, Pain, Function daily living, Function in sports and recreational activities).

SECONDARY OUTCOMES:
Knee function through WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) C scale. | (Day 0, Day 30, Day 90, Day 180 and Day 360)
  To assess knee function through WOMAC C (twelve questions of WOMAC specifically evaluating joint function) scale within 48 hours before the visits. It will be measured the joint function after Hymovis® ONE injection through afive point Likert scale(LK3 series)
Gait analysis system | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation: knee flexion moment, knee flexion angular impulse, knee adduction moment, knee adduction angular impulse
Biomechanical kinematic parameters through gait analysis( tilt at heel contact evaluated per each visit reported | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation tilt at heel contact
Biomechanical kinematic parameters through gait analysis( flexion-evaluated evaluated per each visit reported ) | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation:
  flexion-extension
Biomechanical kinematic parameters through gait analysis(rotation RoM evaluated per each visit reported ) | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation :
  rotation RoM
Biomechanical kinematic parameters through gait analysis(RoM evaluated per each visit reported in the time frame). | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation:
  RoM
Biomechanical kinematic parameters through gait analysis( tilt RoM evaluated per each visit reported in the time frame). | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation:
  tilt RoM
Biomechanical kinematic parameters through gait analysis(flexion-extension evaluated per each visit reported in the time frame). | (Day 0, Day 30, Day 90, Day 180)
  The difference of kinetic parameters will be measured through gait analysis before and after treatment. The following kinetic parameter will be considered for the evaluation :
  flexion-extension
Knee pain through WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) A scale. | (Day 0, Day 30, Day 90, Day 180 and Day 360)
  Knee pain through WOMAC A (five questions of WOMAC specifically evaluating pain) within 48 hours before the visits. It will be measured the knee pain relief after Hymovis® ONE injection through Likert scale
Knee pain through Visual Analogical Scale (VAS, 100 mm, where "No pain = 0" while "Worst Pain Imaginable = 100") | (Day 0, Day 30, Day 90, Day 180 and Day 360)
  Knee pain through Visual Analogical Scale (VAS, 0-100 mm) within 48 hours before the visits. It will be measured the knee pain relief after Hymovis® ONE injection.
The requirement for daily rescue analgesic medication (simple analgesics, acetaminophen) for pain relief. The "rescue dose" will be acetaminophen 3 g per day. | (Day 0, Day 30, Day 90, Day 180 and Day 360)
  The requirement for daily rescue analgesic medication (simple analgesics, acetaminophen) for pain relief. The "rescue dose" will be acetaminophen 3g per day. During the visits patients have to declare the quantity of rescue drug taken and have to deliver at the end of the study the drug left-over
Knee pain, function, stiffness and quality of life through KOOS ((Knee injury and Osteoarthritis Outcome Score) questionnaire. | (Day 0, Day 30, Day 90, Day 180 and Day 360)
  Knee pain and function and quality of life through five items of the KOOS questionnaire. A Likert scale will be used to score each of the five KOOS questionnaire items (Symptoms, Pain, Function daily living, Function in sports and recreational activities). An aggregate score will not be calculated since it is regarded desirable to analyze and interpret the five dimensions separately
The safety of a single i.a. injections by tracking the number of patient withdrawals and their adverse events | (Day 30, Day 60, Day 90, Day 135, Day 180, Day 270 and Day 360)
  The device safety after a single i.a. injection by tracking the number of patient withdrawals and their adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Roma "La Sapienza", Azienda Policlinico Umberto I, Roma, Roma, Italy